CLINICAL TRIAL: NCT02459327
Title: Integrated Model for Promoting Parenting and Early School Readiness in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: University of Pittsburgh (Other); NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1R01HD07639001A1
Record Dates: First submitted 2015-05-26; First posted 2015-06-02 (Estimated); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Infant Behavior; Child Behavior; Parenting; Child Rearing; Depression; Personal Satisfaction; Behavioral Symptoms; Social Control, Informal
Keywords: Infant behavior; Child behavior; Parenting; Child rearing; Depression; Personal satisfaction; Randomized controlled trials; Intervention studies; Behavioral symptoms; Social behavior
MeSH Terms: conditions — Infant Behavior; Child Behavior; Depression; Personal Satisfaction; Behavioral Symptoms; Social Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VIP/FCU (Experimental): VIP (Video Interaction Project) will be offered to all families assigned to the treatment group. FCU (Family Check Up) will be offered to families identified as high risk within the treatment group. Both treatments are parenting interventions.
  Interventions: Behavioral: Video Interaction Project; Behavioral: Family Check Up
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Video Interaction Project — VIP utilizes pediatric well-child visits to build a relationship with an interventionist who facilitates self-reflection regarding interactions with the child through review of videotapes of the parent and child made that day and further facilitates interactions through provision of learning materials (toys and books).
  Other Names: VIP
  Arms: VIP/FCU
Behavioral: Family Check Up — FCU utilizes home visitation to build a relationship with an interventionist who assesses family strengths and challenges and uses motivational interviewing and evidence-based family management strategies to support parent and child behavioral change.
  Other Names: FCU
  Arms: VIP/FCU

SUMMARY:
This study tests a comprehensive approach to the promotion of school readiness in low-income families, beginning shortly after the birth of the child, through enhancement of positive parenting practices (and when present, reduction of psychosocial stressors) within the pediatric primary care platform. The investigators do so by integrating two evidence-based interventions: 1) a universal primary prevention strategy (Video Interaction Project [VIP]); and 2) a targeted secondary/tertiary prevention strategy (Family Check-up [FCU]) for families with infants/toddlers identified as having additional risks. VIP provides parents with a developmental specialist who videotapes the parent and child and coaches the parent on effective parenting practices at each pediatric primary care visit. FCU is a home-based, family-centered intervention that utilizes an initial ecologically-focused assessment to promote motivation for parents to change child-rearing behaviors, with follow-up sessions on parenting and factors that compromise parenting quality.

Two primary care settings serving low-income communities in New York City, NY and Pittsburgh, PA will be utilized to test this integrated intervention in hospital-based clinics, providing information about translation across venues where one of the two interventions has been previously used alone.

The investigators plan to test the VIP/FCU model in a randomized trial of 400 families utilizing parent surveys, observational data on parent-child interactions, and direct assessments of children's development, at key points during intervention follow-up. Analyses will address questions of program impact for the integrated program across all families and by key subgroups.

The largest single contribution made by this study is to test whether an integrated primary and secondary/tertiary prevention strategy implemented in pediatric primary care can produce impacts on early school readiness outcomes, including social-emotional, pre-academic, and self-regulation. As such, this study has the potential to provide the scientific and practice communities with information about an innovative approach to promoting school readiness skills among low-income children.

ELIGIBILITY:
Inclusion Criteria:

* Baby is getting pediatric care at Bellevue Hospital Center or Pittsburgh Children's Hospital
* Caregiver primary language is English or Spanish
* Family can be contacted (has a working phone)
* Family attended second (follow-up) meeting with study team between when the child was aged 10days and 6weeks old

Exclusion Criteria:

* Birth weight <2500gm
* Gestational age < 37 weeks
* Not singleton birth (twin, triplet, etc.)
* Known or suspected significant genetic abnormality
* Known neurodevelopmental/neuromuscular disorder likely to affect development, movement, e.g., seizure disorder, microcephaly (low head circumference)
* Known sensory defect
* Known significant malformation likely to affect development or likely to require significant therapy
* Meets criteria for Early Intervention at birth
* Not in level I nursery at time of enrollment
* Significant postnatal complication requiring level II or III nursery stay. Examples: sepsis, significant hypoglycemia, seizures
* Mother with known significant impairment that will be barrier to communication and participation (e.g., intellectual disability, schizophrenia)
* Baby not being discharged to mother or father
* Mother and baby will be staying in shelter
* Not planning to stay in NYC/ Pittsburgh for at least 3 years
* Has previously participated in VIP or FCU projects
* Baby experiencing significant medical issues
* Doctor has concerns about baby's hearing or vision

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2015-06-03 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Caregiver's cognitive stimulation | When the child is 6 months - 6 years old
  Caregiver's reports of cognitive stimulation. For example engagement in reading, teaching, and play (e.g., StimQ, Dreyer, Mendelsohn, & Tamis-LeMonda, 1995; Mendelsohn, Dreyer, & Tamis-LeMonda, 1999)
Caregiver's harsh parenting and discipline | When the child is 18 months - 6 years old
  Caregiver's reports of discipline strategies (e.g., Socolar et al., 2004; Incredible Years, Webster-Stratton, 2001; Steele et al., 2005)
Caregiver-child interaction quality | When the child is 6 months - 6 years old
  Caregiver's reports and coded videotaped interactions between caregivers and children (e.g., Parenting Young Children, PARYC; McEachern et al., 2011)
Quality of the home environment | When the child is 18 months old
  Observer reports of the home environment (e.g., HOME inventory: Infant-Toddler (IT), Bradley & Caldwell, 1984)
Caregiver depression | When the child is 6 months - 6 years old
  Caregiver's reports of depression (Edinburgh Postnatal Depression Scale (EPDS), Cox, Holden & Sagovsky, 1987; Cox, Chapman, Declan & Jones, 1995)
Caregiver stress/ support | When the child is 6 months - 6 years old
  Caregiver's reports of stress, support, and perceptions of daily hassles (e.g., Abidin Parenting Stress Index, Abidin, 1990; General Life Satisfaction Questionnaire, Crnic, 1983; Parenting Daily Hassle scale, Crnic & Greenberg, 1990; Concern for Children scale, Vines & Baird, 2009)
Child prosocial and problem behavior | When the child is 6 months - 6 years old
  Caregiver's reports of their child's behavioral problems, including externalizing and internalizing problems and prosocial behavior and social skills (e.g., Child Behavior Checklist; Achenbach & Rescorla, 2000; BASC-3, Altmann et al., 2017; Infant-Toddler Social Emotional Assessment, ITSEA, Carter & Briggs-Gowan, 1993; Brief Infant Toddler Social Emotional Assessment, BITSEA, Briggs-Gowan & Carter, 2006; Positive Behavior Scale, Epps et al., 2003)
Children's early language skills | When the child is 6 months - 2 years old
  Caregiver report of non-verbal communication and early expressive language (e.g., MacArthur Communicative Development Inventory; CDI, Fenson et al., 2008; Communication and Symbolic Behavior Scale, CSBS, Wetherby et al., 2001)
Child achievement | When the child is 4 years old - 6 years old
  Direct assessment of children's achievement, including receptive language skills, early academic skills including, reading, math, and writing as well as oral language abilities and academic knowledge (e.g., Receptive One-Word Picture Vocabulary Tests; ROWPVT, Martin and Brownell, 2010; Woodcock Johnson-IV Letter-Word Identification, Applied Problems and Oral Language Comprehension (WJ-IV)/ Bateria III Woodcock-Munoz, Muñoz-Sandoval et al., 2007; McGrew et al., 2014; Test of Word Reading Eficiency (TOWRE), Tarar et al., 2015)
Child executive functioning skills | When the child is 4 years old - 6 years old
  Direct assessment of children's executive functioning, including cognitive skills, inhibitory control, and effortful control (e.g., Dimensional Change Card Sort, DCCS, Zelazo, 2006; Walk a Line, Cookie Waiting, Kochanska et al., 2000)
Caregiver-child relationship quality | When the child is 4 years old - 6 years old
  Caregiver's reports of relationship quality, including the caregiver's perception of conflict and warmth/openness in relationship with the child (e.g., Adult Child Relationship Scale, Pianta & Steinberg, 1991)
Children's self-regulation | When the child is 4 years old - 6 years old
  Observer reports of children's attention/emotional regulation during the direct assessment (e.g., Preschool Self-Regulation Interviewer Assessment, PSRA, Smith-Donald et al., 2007; Moffit Scale, Caspi et al., 1995)

SECONDARY OUTCOMES:
Parenting Quality | Time Frame: When the child is 2 - 4 years old
  Examiner impressions of parenting quality, including measures of responsivity, acceptance, involvement, social skills, and affect. (e.g., items adapted from HOME inventory: Infant-Toddler (IT), Bradley & Caldwell, 1984)
Child temperament | When the child is 6 months, 4 years old, 6 years old
  Caregiver's reports of their child's temperament (e.g., Infant Characteristics Questionnaire, Bates, Freeland, & Lounsbury, 1979; Children's Behavior Questionnaire, CBQ, Rothbart, 2007)
Special services | When the child is 6 months - 6 years old
  Caregiver's reports of their child's Early Intervention referrals and services received
Basic child health | When the child is 6 months - 6 years old
  Attendance in well-child care, growth/ nutrition
Caregiver-child relationship quality | When the child is 18 months - 2 years old
  Caregiver's reports of relationship quality, including the caregiver's perception of conflict and warmth/openness in relationship with the child (e.g., Adult Child Relationship Scale, Pianta & Steinberg, 1991)
Caregiver routines and activities | When the child is 6 months - 6 years old
  Caregiver's reports of routines and activities, including, play, planning, feeding, sleep and media (e.g., McEachern, Dishion, Weaver, Shaw, Wilson, Gardner, 2012; Mendelsohn et al., 2008; Infant Feeding Style Questionnaire, Thompson, A. L., et al. 2009; Parent Teacher Involvement, Kohl et al., 2000)
Caregiver relationship satisfaction | When the child is 6 months - 6 years old
  Caregiver's reports of relationship satisfaction and conflict (e.g., Dyadic Adjustment Scale, Spanier, 1976)
Caregiver regulation of negative emotion | When the child is 24 months old and 6 years old
  Caregiver's reports of their ability to maintain emotional equilibrium when faced with child rearing challenges (e.g., Raver, 2003) and difficulties with emotion regulation (Kaufman et al., 2015)
Caregiver confidence | When the child is 6 months - 4 years old
  Caregiver's reports of their self-efficacy and beliefs related to children's behavior and school readiness. readiness (e.g., adapted Pachter, Sheehan & Cloutier, 2000; Parenting Self-Agency Measure, PSAM, Dumka et al., 1996)
Child narrative comprehension | When the child is 4 years old - 6 years old
  Direct assessment of children's ability to understand and retell narratives, and use higher-order language (e.g., Reese et al., 2012)
Child Theory of Mind | When the child is 4 years old
  Direct assessment of children's ability to mentally represent others' internal states, including measures of false belief and memory control (e.g., Mahy et al., 2017)
Caregiver Mindfulness | When the child is 18 months old
  Caregiver's reports of mindfulness in parenting behavior (e.g., Interpersonal Mindfulness in Parenting, IM-P, Duncan, 2007)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Morris, Ph.D, Principal Investigator — New York University; Alan Mendelsohn, MD, Principal Investigator — NYU Langone Health; Daniel Shaw, Ph.D, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Bellevue Hospital Center, New York, New York
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Mendelsohn AL, Dreyer BP, Flynn V, Tomopoulos S, Rovira I, Tineo W, Pebenito C, Torres C, Torres H, Nixon AF. Use of videotaped interactions during pediatric well-child care to promote child development: a randomized, controlled trial. J Dev Behav Pediatr. 2005 Feb;26(1):34-41. PMID 15718881
- [Background] Shaw DS, Dishion TJ, Supplee L, Gardner F, Arnds K. Randomized trial of a family-centered approach to the prevention of early conduct problems: 2-year effects of the family check-up in early childhood. J Consult Clin Psychol. 2006 Feb;74(1):1-9. doi: 10.1037/0022-006X.74.1.1. PMID 16551138
- [Background] Dishion TJ, Shaw D, Connell A, Gardner F, Weaver C, Wilson M. The family check-up with high-risk indigent families: preventing problem behavior by increasing parents' positive behavior support in early childhood. Child Dev. 2008 Sep-Oct;79(5):1395-414. doi: 10.1111/j.1467-8624.2008.01195.x. PMID 18826532
- [Background] Mendelsohn AL, Huberman HS, Berkule SB, Brockmeyer CA, Morrow LM, Dreyer BP. Primary care strategies for promoting parent-child interactions and school readiness in at-risk families: the Bellevue Project for Early Language, Literacy, and Education Success. Arch Pediatr Adolesc Med. 2011 Jan;165(1):33-41. doi: 10.1001/archpediatrics.2010.254. PMID 21199978
- [Derived] Roby E, Miller EB, Canfield CF, Shaw DS, Morris-Perez PA, Mendelsohn AL. Supporting Early Social-Emotional Competencies Through Reading and Play: Findings From an RCT of the Tiered Smart Beginnings Program. Soc Dev. 2025 Nov;34(4):e70024. doi: 10.1111/sode.70024. Epub 2025 Sep 14. PMID 41394760
- [Derived] Miller EB, Roby E, Zhang Y, Coskun L, Rosas JM, Scott MA, Gutierrez J, Shaw DS, Mendelsohn AL, Morris-Perez PA. Promoting Cognitive Stimulation in Parents Across Infancy and Toddlerhood: A Randomized Clinical Trial. J Pediatr. 2023 Apr;255:159-165.e4. doi: 10.1016/j.jpeds.2022.11.013. Epub 2022 Dec 5. PMID 36481243
- [Derived] Reno R, Whipps M, Wallenborn JT, Demirci J, Bogen DL, Gross RS, Mendelsohn AL, Morris PA, Shaw DS. Housing Insecurity, Housing Conditions, and Breastfeeding Behaviors for Medicaid-Eligible Families in Urban Settings. J Hum Lact. 2022 Nov;38(4):760-770. doi: 10.1177/08903344221108073. Epub 2022 Jul 1. PMID 35775199
- [Derived] Roby E, Miller EB, Shaw DS, Morris P, Gill A, Bogen DL, Rosas J, Canfield CF, Hails KA, Wippick H, Honoroff J, Cates CB, Weisleder A, Chadwick KA, Raak CD, Mendelsohn AL. Improving Parent-Child Interactions in Pediatric Health Care: A Two-Site Randomized Controlled Trial. Pediatrics. 2021 Mar;147(3):e20201799. doi: 10.1542/peds.2020-1799. PMID 33608413
- [Derived] Canfield CF, Miller EB, Shaw DS, Morris P, Alonso A, Mendelsohn AL. Beyond language: Impacts of shared reading on parenting stress and early parent-child relational health. Dev Psychol. 2020 Jul;56(7):1305-1315. doi: 10.1037/dev0000940. Epub 2020 Apr 30. PMID 32352828

DOCUMENTS (1):
  • Informed Consent Form (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT02459327/ICF_000.pdf